CLINICAL TRIAL: NCT06769373
Title: The Effects of Whirlpool Bath and Contrast Bath Treatments on Pain, Disability, Functionality and Grip Strength in Patients with Complex Regional Pain Syndrome After Distal Radius Fracture
Brief Title: The Effects of Whirlpool and Contrast Bath in Patients with Complex Regional Pain Syndrome After Distal Radius Fracture
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Duygu Keskin, Research Assistant Doctor, Afyonkarahisar Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: DK2025
Record Dates: First submitted 2025-01-06; First posted 2025-01-10 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Distal Radius Fracture; Complex Regional Pain Syndrome Type I; Complex Regional Pain Syndrome
Keywords: Whirlpool; Contrast bath; hydrotherapy
MeSH Terms: conditions — Wrist Fractures; Complex Regional Pain Syndromes | interventions — Hydrotherapy

STUDY DESIGN:
Intervention Model Description: Effects of Whirlpool Bath and Contrast Bath Treatments on Pain, Disability, Functionality and Grip Strength in Patients with Complex Regional Pain Syndrome After Distal Radius Fracture. Double-Blinded Prospective Randomized Trial.
Who Masked: Participant, Investigator
Masking Description: Double-Blinded Prospective Randomized Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Whirlpool Bath Protocol (Experimental): An exercise program consisting of hand-wrist range of motion exercises, stretching, strengthening exercises, whirlpool bath therapy and transcutaneous electrical nerve stimulation (TENS) is planned for 4 weeks.
  Interventions: Device: Whirlpool Bath
- Contrast Bath Protocol (Experimental): An exercise program consisting of hand-wrist range of motion exercises, stretching, strengthening exercises, contrasth bath therapy and transcutaneous electrical nerve stimulation (TENS) is planned for 4 weeks.
  Interventions: Device: Contrast Bath

INTERVENTIONS:
Device: Whirlpool Bath — This group of participants will receive an exercise program consisting of 40 minutes hand-wrist range of motion exercises (passive, active assistive), stretching, strengthening exercises, whirlpool bath (32-38 °C) 20 minutes in total, transcutaneous electrical nerve stimulation (TENS) 20 minutes in total for 4 weeks. 5 sessions per week for 20 sessions in the Physical Therapy department.
  Arms: Whirlpool Bath Protocol
Device: Contrast Bath — This group of participants will recieve an exercise program consisting of 40 minutes hand-wrist range of motion exercises (passive, active assistive), stretching, strengthening exercises, contrast bath therapy which consist of 4 minutes hot water (38°C) followed by 1 minute cold water (10°C) periods for 20 minutes in total, transcutaneous electrical nerve stimulation (TENS) 20 minutes in total for 4 weeks. 5 sessions per week for 20 sessions in the Physical Therapy department.
  Arms: Contrast Bath Protocol

SUMMARY:
The aim of our study is to investigate the effects of whirlpool bath and contrast bath treatments on pain, disability, functionality and grip strength in patients with complex regional pain syndrome after distal radius fracture.

DETAILED DESCRIPTION:
Distal radius fractures are the most common fracture type among all body bone fractures. Fractures generally occur in elderly patients caused by low-energy trauma due to decreased bone quality. In young patients, they mostly occur due to traumas such as traffic accidents, falls from heights and sports injuries.

One of the important complications seen after distal radius fractures is complex regional pain syndrome (CRPS). Complex regional pain syndrome represents a complication following distal radius fractures that is still not fully understood etiologically.

Studies have shown that complex regional pain syndrome is commonly diagnosed among patients recovering from a fracture of the distal radius with a reported incidence as high as 37%. It is characterized by excessive pain (allodynia and/or hyperalgesia), edema, local blood flow changes and abnormality of the sudomotor nerve.

There are hardly any studies with a sufficient evidence level to make recommendations for treatments for CRPS-1; therefore, treatment is based on symptom management. Prevention of CRPS-1, after a distal radius fracture is important as this syndrome might lead to chronic pain and serious disabilities. In several studies, it was shown that CRPS-1 can be cured with exercise and graded activities. The main goals of physiotherapy are to reduce pain, regain range of motion, and increase muscle strength and function.

Whirlpool bath and contrast bath treatments are physical therapy methods that has been used safely in complex regional pain syndrome treatment for many years.

Whirlpool baths are local baths where the extremities are immersed in rapidly circulating water. The swirling water produced by the whirlpool bath creates a massaging effect on the body, which can help relieve muscle tension and alleviate pain. The combination of warm water and hydrostatic pressure can also enhance blood circulation and improve joint mobility.

Contrast baths constitute a thermal modality whereby the hand is alternately immersed in hot and cold water for a specified temperature, time, and duration to therapeutically decrease edema, stiffness, pain and increase functionality in cases of complex regional pain syndrome after fractures.

Our primary aim is to investigate the effects of whirlpool bath and contrast bath treatments on pain, disability, functionality and grip strength in patients who were followed conservatively with complex regional pain syndrome (CRPS-1) after distal radius fracture.

ELIGIBILITY:
Inclusion Criteria:

* Patients with complex regional pain syndrome type-1 (CRPS-type 1) after distal radius fracture, who were followed conservatively (long/short arm splint-cast) between the ages of 18-70, who applied to AFSU Physical Medicine and Rehabilitation Clinic. It is planned to use the Budapest diagnostic criteria for the diagnosis of CRPS Type 1.

Exclusion Criteria:

* Orthopedic injuries (other accompanying orthopedic fractures, such as ulna fracture, carpal bone fractures),
* Other system injuries,
* Patients whose distal radius fractures were surgically treated,
* Patients who had previously undergone surgery on the same upper extremity,
* Nerve, tendon and artery injuries accompanying the fracture,
* Other neurological, orthopedic or rheumatological problems affecting the same upper extremity,
* Serious cardiovascular disease,
* Presence of active infection, active dermatitis, skin diseases such as pemphigus, febrile diseases,
* Presence of a fixed catheter in the area,
* Impaired temperature sensationin in the area.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-31 (Estimated); Primary Completion 2025-03-15 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Range of Motion Measurement | up to 12th week
  Supination and pronation of the forearm, flexion, extension, ulnar and radial deviation active/passive range of motion of the wrist will be evaluated with a universal goniometer. Patients will be examined three times in total: before treatment, after treatment (4th week) and at 12th week.
Hand grip strength measurement with Jamar Dynamometer | up to 12th week
  Jamar Dynamometer measures isometric grip force and strength. Measurements will be made by sitting with the shoulder adducted and neutrally rotated, adjacent to the body, elbow flexed at 90 degrees, wrist dorsiflexed at 0-30 degrees and ulnar deviation at 0-15 degrees with the thumb pointing up. Measurements will be repeated three times, 5 seconds apart, on the hand on the affected side, and the average of the three measurements will be recorded in kilograms. Patients will be examined three times in total: before treatment, after treatment (4th week) and at 12th week.

SECONDARY OUTCOMES:
Jebsen Taylor Hand Function Test | up to 12th week
  This test consists of tasks involving types of grasping commonly used in daily life and evaluates the speed of individuals in these tasks.The JTHFT has seven subsets which are writing, simulated page-turning, lifting small objects, simulated feeding, stacking, and lifting large, lightweight, and heavy objects. The test's scoring is recorded as the time it takes for the person to complete the tasks. Patients will be examined three times in total: before treatment, after treatment (4th week) and at 12th week.
The Disabilities of the Arm, Shoulder and Hand Score (Q-DASH) | up to 12th week
  Q-DASH includes 11 items extracted from the DASH questionnaire that measure physical functions and symptoms in patients with upper extremity problems. Each answer is scored from 1 to 5 on a Likert scale from good to bad; 1: no difficulty, 2: mild difficulty, 3: moderate difficulty, 4: extreme difficulty, 5: no ability to do. Each section of the Quick-DASH questionnaire is scored between 0-100 (0= no disability, 100= maximum disability). Patients will be examined three times in total: before treatment, after treatment (4th week) and at 12th week.
Patient-rated Wrist Evaluation Form | up to 12th week
  Patient-rated Wrist Evaluation Form consists of 15 questions that measure the severity of wrist pain and the level of disability in daily life activities. It has two subsections. The pain subsection consists of four questions on pain intensity and frequency, while the function subsection consists of six questions on specific activities and four questions on daily activities. Questions are rated on a 10-point scale (where 0 is no pain and 10 is worst pain). Patients will be examined three times in total: before treatment, after treatment (4th week) and at 12th week.
Short Form 36 (SF-36) | up to 12th week
  SF-36 is a frequently used questionnaire that evaluates the functional health and well-being of patients with 36 different items. These are; physical function, physical role limitation, emotional role limitation, energy/fatigue, mental health, social function, body pain and general health perception. In the evaluation made with this scale, the last 4 weeks are taken into account and the scoring is Likert type except for some items. A total score is calculated separately for each sub-item. The scores are between "0" and "100". While the value of "100" indicates good health status, the value of "0" indicates poor health status. Patients will be examined three times in total: before treatment, after treatment (4th week) and at 12th week.
Visual Analog Scale (VAS) | Up to 12th week
  This method, which is aimed at determining the intensity of pain, aims to have the patient describe their pain with numbers. It is a 10 cm long line that starts with no pain (0) and ends with unbearable pain (10). Patients will be examined three times in total: before treatment, after treatment (4th week) and at 12th week.

CONTACTS AND LOCATIONS:
Locations (1):
- Afyonkarahisar Health Sciences University, Afyonkarahisar, Afyonkarahisar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boersma EZ, Meent HV, Klomp FP, Frolke JM, Nijhuis-van der Sanden MWG, Edwards MJR. Treatment of Distal Radius Fracture: Does Early Activity Postinjury Lead to a Lower Incidence of Complex Regional Pain Syndrome? Hand (N Y). 2022 Jan;17(1):119-127. doi: 10.1177/1558944719895782. Epub 2020 Jan 9. PMID 31916452
- [Background] Jellad A, Salah S, Ben Salah Frih Z. Complex regional pain syndrome type I: incidence and risk factors in patients with fracture of the distal radius. Arch Phys Med Rehabil. 2014 Mar;95(3):487-92. doi: 10.1016/j.apmr.2013.09.012. Epub 2013 Sep 29. PMID 24080349
- [Background] Szekeres M, MacDermid JC, Birmingham T, Grewal R, Lalone E. The Effect of Therapeutic Whirlpool and Hot Packs on Hand Volume During Rehabilitation After Distal Radius Fracture: A Blinded Randomized Controlled Trial. Hand (N Y). 2017 May;12(3):265-271. doi: 10.1177/1558944716661992. Epub 2016 Aug 2. PMID 28453348